CLINICAL TRIAL: NCT03513445
Title: Efficacy of Peri-Incisional Multimodal Drug Injection in Reducing Post-Operative Pain Following Lumbar Spine Surgery
Brief Title: Peri-Incisional Drug Injection in Lumbar Spine Surgery
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORSU-2018-26340
Record Dates: First submitted 2018-04-12; First posted 2018-05-01 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Lumbar Disc Herniation; Degenerative Disc Disease; Spondylolisthesis
MeSH Terms: conditions — Intervertebral Disc Displacement; Intervertebral Disc Degeneration; Spondylolisthesis | interventions — Morphine; Epinephrine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Masking Description: This is a single blind study in which participants are unaware of whether or not they received a peri-incisional injection of pain medication during their surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lumbar Spine Surgery with Injection (Experimental): Patients undergoing lumbar spine surgery will receive a peri-incisional injection of pain medications (morphine, epinephrine, and ropivacaine) during their surgery.
  Interventions: Drug: Morphine; Drug: Epinephrine; Drug: naropin
- Lumbar Spine Surgery without Injection (No Intervention): Patients undergoing lumbar spine surgery will NOT receive a peri-incisional injection of pain medications during their surgery.

INTERVENTIONS:
Drug: Morphine — Morphine, epinephrine, and ropivacaine cocktail will be administered peri-incisionally during lumbar spine surgery.
  Arms: Lumbar Spine Surgery with Injection
Drug: Epinephrine — Morphine, epinephrine, and ropivacaine cocktail will be administered peri-incisionally during lumbar spine surgery.
  Arms: Lumbar Spine Surgery with Injection
Drug: naropin — Morphine, epinephrine, and ropivacaine cocktail will be administered peri-incisionally during lumbar spine surgery.
  Arms: Lumbar Spine Surgery with Injection

SUMMARY:
This is a randomized prospective study that will compare the use of narcotics in a control group of non-injected patients with a treatment arm of patients injected intra-operatively with a ropivacaine, morphine, and epinephrine cocktail. The investigators hypothesize that this treatment will reduce narcotic use in patients during their hospital stay, and possibly decrease the length of their stay in the hospital.The investigators also hope their pain will be decreased as displayed by their multi-daily Clinically Aligned Pain Assessment (CAPA) score.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient 18 years of age and older who is undergoing surgery for a lumbar spine problem. Common diagnoses in this category would include lumbar disc herniations, spinal stenosis, and spondylolisthesis, but this is not an exhaustive list.

Exclusion Criteria:

* Patients with comorbidities excluding use of proposed injection.
* Patients with major head trauma such that they cannot provide consent or describe their post-operative pain.
* Patients with other surgical treatment during study treatment (i.e. more than 1 surgery during the study period or within 30 days prior to surgery).
* Pregnant women (as assessed by pre-operative pregnancy test, which is standard of care).
* Patients with dementia such that they cannot provide consent or describe their post-operative pain.
* Patients with an allergy to study medications.
* Patients with previous drug dependencies.
* Any patient that refuses to be randomized or does not wish to enroll.
* Vulnerable populations, such as prisoners.
* Patients with a fracture, tumor, or infection as their primary diagnosis.
* Patients undergoing a deformity correction.
* Patients with surgeries extending more than 4 levels, with surgeries that extend to the pelvis, or with surgeries that cross the thoracolumbar junction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Post-operative narcotic use | Up to 6 weeks

SECONDARY OUTCOMES:
Patients' self-reported pain (CAPA) scores | Up to 6 weeks
  Evaluates
  * intensity of pain
  * effect of pain on functionality
  * effect of pain on sleep
  * efficacy of therapy
  * progress toward comfort
Length of hospital stay | Up to 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No